CLINICAL TRIAL: NCT04100395
Title: Global Hemostasis Monitoring in Patients With Severe Trauma Using Sonoclot Signature Compared to Conventional Coagulation and Platelet Parameters
Brief Title: Global Hemostasis Monitoring by Using Sonoclot Signature in Traumatic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, DO Ahmed, Resident physician, Assiut University
Other Study IDs: sonoclot signature
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Study of Hemostatic Profile in Traumatic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sonoclot — Sonoclot Analyzer is best described as a microviscometer. The electronics are sensitive to any resistance to motion that the oscillating probe encounters as it moves within the test sample.

SUMMARY:
1. Analyzing the effects of severe trauma using sonoclot analyzer (which depicts the entire hemostatic pathway) ,subsequently describing the convenient therapy .
2. Assessing the correlations between sonoclot variables and conventional coagulation and platelet function tests

DETAILED DESCRIPTION:
Coagulopathy is a physiological response to massive bleeding that frequently occurs after severe trauma and is an independent predictive factor for mortality[2]. . There are two of the major causes of coagulopathy in trauma patients

1. coagulopathy secondary to hemorrhagic shock due to massive bleeding and
2. coagulopathy secondary to severe head injury[3] which results in release of tissue factor from damaged brain tissue.

Therefore, it is very important to grasp the coagulation status of patients with severe trauma quickly and accurately with objective indicator in order to establish the therapeutic strategy .

The importance of viscoelastic devices in understanding the disease condition of patients with traumatic coagulopathy has been widely recognized in Europe. Viscoelastic hemostatic assays devices have practical advantages as point-of-care devices for monitoring major hemorrhage including speed of results and a set of parameters that assesses a global coagulation profile .

Also In the USA, Massive Transfusion in Trauma Guidelines proposed by the American College of Surgeons in 2013 presented the test results obtained by the viscoelastic devices, as the standard for transfusion or injection of blood plasma, cryoprecipitate, platelet concentrate, or anti-fibrinolytic agents in the treatment strategy for traumatic coagulopathy and hemorrhagic shock .

However, some studies have reported limitations of these viscoelastic devices

ELIGIBILITY:
Inclusion Criteria:

* -Patients >18 years.
* Both sexes will be included.
* Recent trauma

Exclusion Criteria:

* -patients <18 years.
* Patients with documented evidence of coagulopathy or bleeding diocese .
* Patients with liver disease.
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study will be done on patients sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2032-10-15 (Estimated)

PRIMARY OUTCOMES:
global monitoring of coagulation profile | baseline
  Viscoelastic hemostatic assays devices have practical advantages as point-of-care devices for monitoring major hemorrhage including speed of results and a set of parameters that assesses a global coagulation profile